CLINICAL TRIAL: NCT02172118
Title: Pharmacokinetics, Safety and Tolerability of Single Dose of BI 1744 CL (30 μg Administered With the Respimat® Inhaler) in Patients With Severe Renal Impairment in Comparison to Subjects With Normal Renal Function in a Monocentric, Open Label, Parallel Group Phase I Trial
Brief Title: BI 1744 CL in Patients With Severe Renal Impairment in Comparison to Subjects With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1222.35
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (2):
- severely renally impaired patients (Experimental)
  Interventions: Drug: BI 1774 CL
- healthy volunteers (Experimental)
  Interventions: Drug: BI 1774 CL

INTERVENTIONS:
Drug: BI 1774 CL

SUMMARY:
Study to assess the influence of severe renal impairment on the pharmacokinetics (PK), safety, and selected pharmacodynamic (PD) parameters of BI 1744 CL (30 μg administered by inhalation with the Respimat® Inhaler)

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects:

* Healthy male and female subjects determined by results of screening with a creatinine clearance >80 mL/min (Treatment Group 2)
* Age 21 - 75 years
* Body Mass Index (BMI) >=18.5 and <=32 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Renally impaired subjects:

* Renally impaired male or female subjects (Treatment Group 1) determined by results of screening with the following creatinine clearance as estimated according to Cockroft-Gault: Creatinine clearance <30 mL/min (Treatment Group 1, Renal Function Group 4)
* Age 21 - 75 years
* BMI >=18.5 and <=34 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion Criteria:

Healthy subjects who meet any of the following criteria will not be entered into this trial:

* Any finding of the medical examination (including blood pressure (BP) [>140 mmHg systolic and or >95 mmHg diastolic], pulse rate (PR) and electrocardiogram (ECG)) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Relevant gastrointestinal tract surgery (except appendectomy, herniotomy)
* Diseases of the central nervous system (such as epilepsy, seizures) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections (e.g. including Hepatitis B and C and HIV)
* History of allergy/hypersensitivity (including drug allergies) that are deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Participation in another trial with an investigational drug within one month after previous single dose administration or two months after previous multiple dose administration prior to administration or during the trial
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking when confined to the study site on trial days
* Alcohol abuse (more than 40 g/day in males, more than 20 g/day in females)
* Drug abuse, in the investigator's judgement upon review of the patient's history and urine screening for abused substances
* Veins unsuited for iv puncture on either arm (e.g. veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture)
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within 48 hours prior to trial or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of study centre
* Subjects not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions

Renally impaired subjects who meet any of the following criteria will not be entered into this trial:

* Moderate and severe concurrent liver function impairment (e.g. due to hepatorenal syndrome)
* Patients with significant diseases other than renal impairment will be excluded. A significant disease is defined as a disease which in the opinion of the investigator

  * put the patient at risk because of participation in the study
  * may influence the results of the study
  * may influence the patient's ability to participate in the study
  * is not in a stable condition

    * Diabetic or hypertensive patients can be entered in this trial if the disease is not significant according to these criteria.
* Relevant gastrointestinal tract surgery (except appendectomy, herniotomy)
* Diseases of the central nervous system (such as epilepsy, seizures) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections (e.g. including Hepatitis B and C and HIV)
* History of allergy/hypersensitivity (including drug allergies) that are deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial, excluded are those drugs, the patient is currently taking for treatment of the renal or concomitant disease
* Subjects with a change of their chronic medication less than 4 weeks prior to dosing
* Participation in another trial with an investigational drug within one month after previous single dose administration or two months after previous multiple dose administration prior to administration or during the trial
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking when confined to the study site on trial days
* Alcohol abuse (more than 40 g/day in males, more than 20 g/day in females)
* Drug abuse, in the investigator's judgement upon review of the patient's history and urine screening for abused substances
* Veins unsuited for iv puncture on either arm (e.g. veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture)
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within 48 hours prior to trial or during the trial)
* Clinically relevant laboratory abnormalities (except for renal function tests or deviations of clinical laboratory values that are related to renal impairment)
* Hemoglobin < 8 g/dL indicating severe renal anemia (use of erythropoetin is allowed to maintain hematocrit)
* Inability to comply with dietary regimen of study centre
* Subjects not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions
* Systolic blood pressure < 100 or > 180 mm Hg, diastolic blood pressure < 60 or > 110 mm Hg, pulse rate < 50 or > 100 1/min

Exclusion criteria specific for this study due to the known class side effect profile of ß2- mimetics (healthy or renally impaired subjects):

* Asthma or history of pulmonary hyperreactivity
* Hyperthyrosis
* Allergic rhinitis in need of treatment
* Clinically relevant cardiac arrhythmia

For female subjects (healthy or renally impaired):

* Pregnancy or planning to become pregnant within 2 months of study completion
* Positive pregnancy test
* No adequate contraception in women of childbearing potential (adequate contraception: e.g. sterilisation, intrauterine device or oral contraception not containing ethinyl estradiol or ethinyl estradiol with an additional barrier method) for at least 3 months prior to participation in the study
* Inability to maintain this adequate contraception during the whole trial period
* Lactation period

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
AUC0-4 (area under the concentration time curve of the analyte in plasma over the time interval from 0 to 4 hours after dosing) | before and at 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, 72:00 hours following drug administration
Cmax (maximum concentration of the analyte in plasma) | before and at 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, 72:00 hours following drug administration

SECONDARY OUTCOMES:
tmax (time from dosing to the maximum concentration of the analyte in plasma) | before and at 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, 72:00 hours following drug administration
AUC (area under the concentration-time curve of the analyte in plasma at different time points) | before and at 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, 72:00 hours following drug administration
%AUCtz-∞ (percentage of area under the concentration-time curve obtained by extrapolation) | before and at 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, 72:00 hours following drug administration
λz (terminal rate constant in plasma) | before and at 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, 72:00 hours following drug administration
t1/2 (terminal half-life of the analyte in plasma) | before and at 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, 72:00 hours following drug administration
MRTih (mean residence time of the analyte in the body after inhalation) | before and at 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, 72:00 hours following drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | before and at 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, 72:00 hours following drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | before and at 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, 72:00 hours following drug administration
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to t2) | before and at 0-8, 8-12, 12-24, 24-48, 48-72 hours following drug administration
fet1-t2 (fraction of analyte excreted in urine from the time point t1 to t2) | before and at 0-8, 8-12, 12-24, 24-48, 48-72 hours following drug administration
CLR,t1-t2 (renal clearance of the analyte in plasma from the time point t1 to t2) | before and at 0-8, 8-12, 12-24, 24-48, 48-72 hours following drug administration
Plasma protein binding of BI 1744 BS | before and at 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, 72:00 hours following drug administration
Number of patients with adverse events | up to 5 weeks
Assessment of tolerability on a 4-point scale by the investigator | within 5 to 14 days after drug administration